CLINICAL TRIAL: NCT02280005
Title: First 24 Hour Human Trial of the Wearable Artificial Kidney
Brief Title: 24 Hour Use of the Wearable Artificial Kidney
Acronym: WAK US 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blood Purification Technologies, Inc. (Industry)
Collaborators: University of Washington (Other); Wearable Artificial Kidney Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WAK Seattle
Record Dates: First submitted 2014-09-19; First posted 2014-10-31 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: End Stage Renal Disease
Keywords: Dialysis; Renal Failure; Wearable; Artificial Kidney; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WAK Treatment (Experimental): Use of experimental device.
  Interventions: Device: WAK Treatment

INTERVENTIONS:
Device: WAK Treatment — Hemodialysis with WAK device.

SUMMARY:
This is a prospective, interventional study designed to provide preliminary data on the human use of the WAK. Up to 10 subjects currently receiving intermittent hemodialysis (HD) treatment three times per week for end-stage renal disease (ESRD) via an indwelling tunneled catheter will be studied.

DETAILED DESCRIPTION:
Subjects will undergo 24 hours in-hospital treatment with the Wearable Artificial Kidney (WAK). Up to 10 subjects with ESRD will complete the protocol in its entirety.

The objective of this protocol is to provide additional preliminary data supporting the hypothesis that the WAK safely and effectively delivers dialysis therapy that is at least equal to the current standard of care for treatment of ESRD using conventional machines for thrice weekly hemodialysis treatments. These objectives would be accomplished by absence of adverse events during treatment with the WAK, along with effective removal of fluid and solutes at least equal to those delivered with conventional currently used dialysis machines. The WAK will be the only investigational device used in this study.

The reason for this trial is to advance the eventual approval of this device to be legally commercialized as it potentially may respond to the unmet public health needs to improve outcomes and reduce costs in the treatment of ESRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and competent to sign the approved informed consent.
* Patient must be at least 21 years of age or older.*
* Patient must weigh between 45 and 100kg, inclusive.*
* Patient must have End Stage Renal Disease and currently undergoing consistent intermittent HD at least 3 times a week for at least 3 months prior to being enrolled.*
* Vascular access must be through a functioning double lumen catheter with no thrombolytic therapy or clotting of the catheter within the past 4 weeks.*
* Willing to comply with the requirements of experimental treatment with the WAK for up to 24 hours.
* Expected survival of no less than 6 months.*
* Consent to allow review of their medical records by the investigators, and monitors.
* Fluency in English
* Hemoglobin level ≥ 9.0 g/dL prior to WAK treatment

Exclusion Criteria:

* • Anticipating or scheduled for a living related donor kidney transplant in less than 2 months.**

  * History (within the 12 weeks prior to the study) of cardiovascular events including:*

    * Unstable angina
    * Myocardial Infarction
    * Stroke
    * Clinical Significant Arrhythmia
  * Life threatening arrhythmia within the past 30 days*
  * Severe intradialytic hypotension within the last 30 days*
  * Shock within the last 30 days*
  * Hemodynamic instability as demonstrated by repeated episodes of hypotension or hypertension requiring intervention by dialysis personnel or representing a present hazard to the patient*
  * Seizure disorder requiring active treatment for a seizure episode during the last 6 months*
  * Major Surgery (excluding vascular access surgery) within the past 30 days *
  * Currently receiving intravenous antibiotic therapy for systemic infection*
  * Clinical evidence of metastatic malignancy, receiving radiation or chemotherapy, within the past 365 days*
  * Active bleeding*
  * Hematological disease (e.g. malignancies, hemolytic anemia, thrombocytopenia), and other conditions that may interfere of confuse the data obtained from this trial.*
  * Current enrollment in another investigational device or drug trial.**
  * Subject is pregnant (e.g., positive HCG test) or is breast feeding.
  * Subject has any disorder (excluding illiteracy or visual impairment) that compromises the ability of the subject to give written informed consent and/or to comply with the study procedures.*
  * Allergy to heparin or ethylene oxide.*
  * Hypertension deemed uncontrolled, at the discretion of the investigator, within the past 30 days.*
  * Has an implantable electronic device (e.g. pacemaker)*

    * As documented in patient medical history (see attached). **Patient self-report.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours
Subject vital signs as a Measure of Safety and Tolerability | 24 hours
Satisfaction survey as a Measure of Safety and Tolerability | Post Treatment
Blood creatinine as a Measure of Safety and Tolerability | 24 hours
Dialysate toxin load as a Measure of Safety and Tolerability | 24 hours
Blood electrolytes as a Measure of Safety and Tolerability | 24 Hours

SECONDARY OUTCOMES:
Blood urea levels | 24 hours
Dialysate Urea Levels | 24 hours
Blood creatinine levels | 24 hours
Dialysate creatinine levels | 24 Hours
Volume of spent dialysate | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Gura V, Rivara MB, Bieber S, Munshi R, Smith NC, Linke L, Kundzins J, Beizai M, Ezon C, Kessler L, Himmelfarb J. A wearable artificial kidney for patients with end-stage renal disease. JCI Insight. 2016 Jun 2;1(8):e86397. doi: 10.1172/jci.insight.86397. PMID 27398407